CLINICAL TRIAL: NCT00184977
Title: A Double-blind Placebo-controlled Trial Comparing the Efficacy and Cost-effectiveness of Inhaled Fluticason Propionate Versus Oral N-acetylcysteine in the Treatment of Patients With COPD in General Practice
Brief Title: COPD on Primary Care Treatment (COOPT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Health Care Insurance Board (CVZ) (Unknown); GlaxoSmithKline (Industry); Zambon SpA (Industry); The Netherlands Asthma Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 98-46140; 95093 FLU9802 NAC-NL-11
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2010-03-12 (Estimated); Status verified 2006-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive; Bronchitis, Chronic
Keywords: Pulmonary Disease, Chronic Obstructive; Randomized Controlled Trial; Family Practice; Respiratory Function Tests; Health Status
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive; Bronchitis, Chronic | interventions — Acetylcysteine; Fluticasone

INTERVENTIONS:
Drug: N-acetylcysteine
Drug: fluticasone propionate

SUMMARY:
The aim of this family practice based study is to determine the long-term treatment effects of two drugs that are presumed to modify the course and progression of chronic obstructive pulmonary disease (COPD), oral N-acetylcysteine and inhaled corticosteroids.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a disorder characterised by symptoms and abnormal tests of expiratory flow that do not change markedly over periods of several months observation. COPD includes chronic bronchitis and emphysema. It is not fully clear which medication is the most efficacious in the long-term treatment of COPD. In contrast to asthma, the efficacy and therefore the precise role of inhaled corticosteroids is less clear in the treatment of patients with COPD. The same applies to another (much less investigated) possibility in the treatment of COPD, the anti-oxidant agent N-acetylcysteine. N-acetylcysteine is used as a mucolytic agent in a variety of clinical conditions, such as acute and chronic bronchitis and cystic fibrosis. The aim of this study, which is performed in family practices, is to determine the 3-year treatment effects and cost-effectiveness of oral N-acetylcysteine versus an inhaled corticosteroid (fluticason propionate) in modifying the course and progression of COPD.

Comparisons: N-acetylcysteine (oral, 600 mg o.d.) and fluticason propionate (dry powder inhalation, 500 mcg b.i.d.) are compared with placebo

ELIGIBILITY:
Inclusion Criteria:

* age between 30 and 75 years
* being a smoker or ex-smoker
* post-bronchodilator FEV1/FVC ratio is <88% of the predicted value in case of men or <89% of the predicted value in case of women
* post-bronchodilator FEV1>=40% and <90% of the predicted value
* subjects have a GP diagnosis of COPD or had increased cough, sputum and/or dyspnea on most days for 3 or more months a year, for at least the last 2 years
* able to provide a written informed consent
* expected to be able to comply with the study protocol
* able to communicate with the study personnel and to understand and read instructions
* females of childbearing potential should use an acceptable method for birth control

Exclusion Criteria:

* a known history of intolerance or allergy for N-acetylcysteine or fluticason
* use of long-term oxygen therapy or expected to be in need of oxygen therapy within the next 3 years
* registered asthma, allergic rhinitis, and/or allergic eczema as an active problem in the GPs records within the last 12 months
* alpha1-antitrypsin deficiency
* cystic fibrosis
* active infection due to Mycobacterium tuberculosis
* status post-lobectomy
* clinically proven gastric or duodenal ulcer in the previous six months
* non-compensated severe chronic congestive heart failure
* life expectancy reduction (e.g. malignancies)
* evidence of illicit drug use or abuse of alcohol intake
* expected not to be compliant in taking medications in general
* being pregnant or giving breastfeeding
* not complying with the inclusion criteria

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270
Dates: Start 1998-12; Study Completion 2003-01

PRIMARY OUTCOMES:
exacerbations of COPD, condition-specific quality of life

SECONDARY OUTCOMES:
lung function decline, respiratory symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Tjard RJ Schermer, MSc, PhD, Principal Investigator — Radboud University Nijmegen Medical Centre, Department of Family Medicine; Chris van Weel, MD, PhD, Study Director — Radboud University Nijmegen Medical Centre, Department of Family Medicine
Locations (2):
- Netherlands (2):
  - Department of Family Medicine, University of Maastricht, Maastricht
  - Department of Family Medicine, Radboud University Nijmegen Medical Centre, Nijmegen

REFERENCES:
- See also: Department of General Practice/Family Medicine, Radboud University Nijmegen Medical Centre — http://www.umcn.nl/Pages/default.aspx
- See also: Health Care Insurance Board (CVZ) — http://www.cvz.nl/
- See also: Netherlands Asthma Foundation — http://www.astmafonds.nl
- See also: Dutch Health Care Inspectorate — http://www.igz.nl
- See also: GlaxoSmithKline (study sponsor) — http://www.gsk.com
- See also: Zambon Group Spa (Study Sponsor) — http://www.zambongroup.com